CLINICAL TRIAL: NCT05967026
Title: Characterization of Myocardial Infarction Scar Using Magnetic Resonance Imaging
Acronym: MI-SCAR-MRI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, HAMMACHE Nefissa, Residant in Cardiology Unit, Central Hospital, Nancy, France
Other Study IDs: 2023PI071
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Myocardial Infarction
Keywords: cardiac magnetic resonance; sudden cardiac death; risk stratification
MeSH Terms: conditions — Myocardial Infarction; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this monocentric observationnal study is to describe the characteristics of the myocardial infarction scar in terms of transmurality in residual LVEF>35% patients.

The primary objective is to determine the frequency of the criterion "intramural scar ≥1.47cm2" (measured by MRI) in patients who presented with myocardial infarction with residual LVEF≥35%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ;
* History of acute coronary syndrome prior to inclusion and having undergone cardiac MRI;
* LVEF >35% measured at least 6 weeks post-IDM by echocardiography or MRI;

Exclusion Criteria:

- Patient with an implantable cardiac device (implantable cardioverter defibrillator or pacemaker) prior to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a history of acute coronary syndrome prior to inclusion and having undergone cardiac MRI and LVEF >35% measured at least 6 weeks post-IDM by echocardiography or MRI
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Intramural scar surface in cm² | 6 weeks after myocardial infarction
  Intramural scar surface in cm²>1.47cm²

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Nancy, Nancy, France